CLINICAL TRIAL: NCT02649595
Title: Bridge Copenhagen - Respite Care for Homeless People
Acronym: BC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Red Cross Copenhagen (Unknown); Region Capital Denmark (Other); Copenhagen Municipality, Denmark (Other Government)
Responsible Party: Principal Investigator, Ove Andersen, Research Director, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15000708; 04173 AHH-2015-090 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Homelessness; Respite Care
Keywords: Homeless; Homelessness; Respite care; EQ-5D; Quality of life questionnaire; Economic evaluation; Cost-utility analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red Cross respite care (Other): A 2 week free stay at a Red Cross respite center after hospitalization.
  Interventions: Other: Red Cross Respite care
- Streets/communal programmes (No Intervention): Homeless being discharged from hospital to the streets and communal programmes.

INTERVENTIONS:
Other: Red Cross Respite care — See detailed description.
  Other Names: Omsorgscenter Thorsgade
  Arms: Red Cross respite care

SUMMARY:
The aim of this study is to determine the effect of a two week respite program (Red Cross) for homeless people just discharged from hospitals in the capital region of Denmark.

The study is a randomized controlled trial and an economic evaluation. The intervention is a 2 week stay at a Red Cross respite care center. The intervention is intended for homeless people or functional homeless, who has been admitted to hospital and received standard medical care and treatment at the hospital. Under normal circumstances the homeless patients would be discharged to live on the street and receive care from programs in the municipalities. The respite center offers standard nursing care, rest with a place to sleep, food and help dealing with social problems such as economy and housing. The respite care center is led by a nurse who is represented during daytime from Monday to Friday and besides that, volunteers are used as staff.

The control group is receiving usual care and is discharged to the street and the usual communal programs.

The study examines whether a 2 week stay is cost effective and whether it can improve the health related quality of live (HRQoL). The hypothesis is that a respite care stay will result in a 25 % reduction in health care costs and increase the HRQoL.

DETAILED DESCRIPTION:
The study is a randomized controlled trial with an economic evaluation of a Red Cross respite care stay for homeless people, who have just been discharged from hospital in the capitol region of Denmark.

The effect of a respite care stay for homeless people has never been investigated in Denmark.

Intervention:

The intervention consists of a 2 week stay at a Red Cross respite center. The intervention is intended for homeless or the functional homeless who is not ill enough to stay in the hospital, but to sick or frail to live on the streets. The homeless patients have received the standard medical care and treatment at the hospital and would under normal circumstances be discharged to live on the street and receive care from programs in the municipalities. The respite care center offers a free stay with a place to sleep, food three times a day, help with nursing tasks and help dealing with social problems such as economy and housing. The place is led by a nurse who is working during daytime from Monday to Friday and besides that, volunteers are used as staff.

The control group is discharged from hospital to the street and the usual programs in the municipalities.

Outcome:

The primary outcome is the difference in health economic costs measured in DKK over a period of 3 months. The secondary outcomes are difference in Quality adjusted life-years (QALY) over a period of 3 month, health economic costs over a period of 6 months, difference in elective health care costs, difference in acute health care costs and difference in social costs.

Quality adjusted life-years can be calculated by using the EQ-5D-5l questionnaire that measures health related quality of life (HRQoL). The answers from the questionnaire can be converted to an index value and is used to calculate QALY's. Quality Adjusted Life-Years is also used as the outcome measure of the cost-utility analysis (CUA).

Data collection:

Data about health economic costs for the CUA is going to be extracted from the National Patient Registry, Civil Registration System, The National Health Insurance Service Registry, communal databases and from the operational costs of the respite center.

HRQoL is measured by using the questionnaire EQ-5D-5L. All participants answer the questionnaire at baseline at the hospital before randomization, then 2 weeks later and again 3 month from baseline. The answers from the questionnaire can be converted to an index value and is used to calculate Quality Adjusted Life-years (QALY). In this way it can be investigated whether there has been an increase or decrease in QALY's and clarify if there is any difference between the two groups.

Variables:

There will be collected information on following variables, demographics, mental illness (reported from latest hospital admission by the social nurses), physical health by Charlson score, self-reported substance abuse and duration of homelessness. Moreover records from the Red Cross respite center will be reviewed and information about what the individuals received help with is registered.

Analyses:

Regarding the primary outcome, an analysis of variance is performed to determine the difference between the costs of the intervention and control group. Furthermore analysis of variance is performed to compare the development in QALY's in both groups. Both the analysis for the primary and secondary outcome is performed as an intention to treat analysis.

The economic evaluation is performed like a CUA. Results from the CUA will be presented as an incremental cost-effectiveness ratio (ICER).

In case of a skew distribution between intervention and control group in possible confounders like the variables mentioned above, the analysis will also be adjusted for these.

Sample size:

With a power of 80 %, p- values=0,05, an estimated health economic costs in the control group on 100.000 DKK and a standard deviation of 39.243 DKK. To detect a difference between the groups of minimum 25.000 DKK, a total of 96 participants are needed in the study. That includes 20 % drop-out for data regarding the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Homeless or functional homeless who is self-reliant and not ill enough to stay in the hospital but to sick or frail to live on the streets.

Exclusion Criteria:

* People who has cognitive problems understanding the information about the study.
* People who does not speak and understands at least one of the following languages: Danish, english, polish, romanian, german and french.
* People who have planned to leave Denmark within 6 month of inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Health economic costs | 3 months
  All costs related to health extracted from the National Patient Registry, Civil Registration System, The National Health Insurance Service Registry, databases from the municipality and from information about costs from the Red Cross respite center. Hereby it can be investigatet if there is any difference in health economic costs between the two groups.

SECONDARY OUTCOMES:
Health Related Quality of Life (EQ-5D-5L) | 3 months
  HRQoL is measured by using the questionnaire EQ-5D-5L. All participants answer the questionnaire at baseline at the hospital, 2 weeks later and again 3 month from baseline. The answers from the questionnaire can be converted to an index value and is used to calculate Quality Adjusted Life-years (QALY). In this way it can be investigated if there is difference in QALY's between the two groups.
Health economic costs | 6 months
  All costs related to health extracted from the National Patient Registry, Civil Registration System, The National Health Insurance Service Registry, databases from the municipality and from information about the budget of the Red Cross respite center. Hereby it can be investigatet if there is any difference in health economic costs between the two groups.
Elective health care costs | 3 and 6 months
  Data on elective health costs will be retrieved from the National Patient Registry, The National Health Insurance Service Registry and databases from the municipalities to see if there is a difference between the control group and the intervention group
Acute health care costs | 3 and 6 months
  Data on acute health care costs will be retrieved from the National Patient Registry, The National Health Insurance Service Registry and databases from the municipalities to see if there is a difference between the control group and the intervention group
Social costs | 3 and 6 months
  Data on social costs will be retrieved from the National Patient Registry, The National Health Insurance Service Registry and databases from the municipalities to see if there is a difference between the control group and the intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, PhD, MD, Principal Investigator — Clinical Research Centre, University Hospital of Copenhagen, Hvidovre
Locations (1):
- Clinical research Centre, Amager Hvidovre hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Bring C, Kruse M, Ankarfeldt MZ, Brunes N, Pedersen M, Petersen J, Andersen O. Post-hospital medical respite care for homeless people in Denmark: a randomized controlled trial and cost-utility analysis. BMC Health Serv Res. 2020 Jun 5;20(1):508. doi: 10.1186/s12913-020-05358-4. PMID 32503545